CLINICAL TRIAL: NCT01113788
Title: Tricuspid Isthmus Architecture as Imaged by CARTOsound, Determines Ablation Times in Patients With Typical Atrial Flutter
Brief Title: Tricuspid Isthmus Imaged by CARTOsound, Patients With Typical Atrial Flutter
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Dr. Allan Skanes, UWO Department of Medicine
Other Study IDs: R-09-414; 16214 (Other: REB)
Record Dates: First submitted 2010-01-11; First posted 2010-04-30 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Atrial Flutter
Keywords: atrial flutter, tricuspid isthmus, ablation
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- imaging: imaging with usual catheter/fluoroscopy, no cartosound
  Interventions: Device: tricuspid isthmus imaging with Cartosound

INTERVENTIONS:
Device: tricuspid isthmus imaging with Cartosound — tricuspid isthmus imaging with Cartosound
  Other Names: Cartosound

SUMMARY:
The investigators propose a third hypothesis based on the anatomic observations made in pathological studies. The investigators hypothesize that the anatomic architecture determines the functional properties of the TV-IVC isthmus. As a result,

• Muscular bundles are preferential routes of conduction through the TV-IVC isthmus. The isthmus acts like a series of discreet conduction routes rather than as a sheet of tissue.

The muscular bundles form selective targets for ablation and therefore the entire anatomic line need not be ablated. This has direct implications for ablation of the isthmus.

DETAILED DESCRIPTION:
Patients undergoing atrial flutter ablation will have cartosound imaging done during procedure to determine if this will shorten ablation times.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over 18 years of age provided written informed consent documented atrial flutter by ECG , holter monitor or TTM

Exclusion Criteria:

* previous atrial flutter ablation non isthmus dependent atrial flutter prior right atrial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with typical atrial flutter
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
observational including ablation lesion number, ablation time in minutes, fluoroscopic | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan Skanes, MD, FRCPC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Center, London, Ontario, Canada